CLINICAL TRIAL: NCT04454216
Title: GSD VI and GSD IX Natural History
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00104116
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Glycogen Storage Disease VI; GLYCOGEN STORAGE DISEASE IXa1; GLYCOGEN STORAGE DISEASE IXa2; Glycogen Storage Disease IXB; Glycogen Storage Disease IXC; GSD 9 (All Subtypes); GSD 6
MeSH Terms: conditions — Glycogen Storage Disease Type VI; Glycogen Storage Disease, Type IXA2; Glycogen Storage Disease IXB; Glycogen Storage Disease IXC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is an observational study that consists of data abstraction from patient medical records.

SUMMARY:
Collection and review of clinical information related to Glycogen Storage Disease Type VI (GSD VI) OR Glycogen Storage Disease Type IX (GSD IX) generated during clinic visits.

DETAILED DESCRIPTION:
This natural history study will serve as a repository of clinical, laboratory, and biochemical information on individuals with GSD VI or GSD IX. This information will allow a more definitive description of glycogen phosphorylase (GP) and phosphorylase kinase (PhK) deficiency to be developed, which will permit development of treatment strategies for these diseases.

Duke will be the only site where this study takes place. However, since these are rare disorders, participants who receive care at other institutions will be included. The investigators will collect retrospective data from patient charts on diagnosed individuals, as far back as necessary to capture the clinical course of the disorder. Prospective data collected from patient charts after enrollment will be captured as well. Participant's medical records will be continually reviewed for the duration of the study.

Data will be collected from medical records and will only pertain to clinically relevant information, including, but not limited to: demographic and diagnostic information, tissue biopsy results, medical and family history, review of systems, imaging studies, results of liver and/or muscle testing, and urine and blood laboratory results.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GSD VI or GSD IX via:

  * Two variants in the PYGL, PHKA1, PHKA2, PHKG1, PHKG2, or PHKB gene (or one variant with evidence of disease). Note: for males, one variant in the PHKA1 or PHKA2 gene is sufficient for inclusion.
  * Deficient GP activity or PhK activity per enzymology
  * Histology as confirmed by clinician
* Pregnant women with a diagnosis of GSD VI or GSD IX will be included
* Able to provide informed consent for self (adults) or affected individual (minor or adults with a legally authorized representative)
* Able to provide consent for release of medical records

Exclusion criteria:

* Unable to provide informed consent for participation for one's self or by legally authorized representative/legal guardian/parent

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with GSD VI or GSD IX, regardless of gender or ethnicity, are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression of disease confirmed by medical record review | through study completion, an average of 10 years
Serum biotinidase activity | through study completion, an average of 10 years
Number of genotypes presented | through study completion, an average of 10 years
Number of phenotypes presented | through study completion, an average of 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kishnani, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koch RL, Fares AH, Cocanougher BT, Lim J, Haijer-Schreuder AB, Derks TGJ, Grunert SC, Sharma R, Jones KA, Kishnani PS. PHKA1-associated phosphorylase kinase deficiency: a monogenic disorder of exercise intolerance and myalgia. NPJ Genom Med. 2025 Nov 10;10(1):71. doi: 10.1038/s41525-025-00527-y. PMID 41213961